CLINICAL TRIAL: NCT03453879
Title: TeamOBS - Focuses on the Association Between Teamwork and Clinical Performance in Emergency Obstetrical Situations
Brief Title: Observation of Emergency Obstetrical Situations.
Acronym: TeamOBS
Status: Completed | Type: Observational
Sponsor: TeamOBS (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Horsens Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2016-04-12; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Unspecified Obstetrical Trauma, With Delivery; Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Study population: Participants in this study are working staff (junior and senior doctors, midwifes and other health personal) in the maternity wards of two hospitals in Central Region Denmark: Horsens Regional Hospital and Aarhus University Hospital, Skejby.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention - only observation of teams delivering acute obstetric care

SUMMARY:
The TeamOBS study is an observational study. We analyze actually recordings of obstetric emergencies to get an even better understanding and knowledge of the association between the communication and cooperation and the quality of the performance of the interdisciplinary team.

DETAILED DESCRIPTION:
Background:

In obstetric emergency situations (OES) inadequate non-technical skills (NTS) are the leading causes of substandard care.

Aim:

Based on live audio and video (AV)-recordings of real (OES) the aim is to describes how the NTS and the clinical performance are related.

Method:

1. Inclusion of the teams. OES teams from the delivery ward at two Danish hospitals, Aarhus University Hospital and Horsens Regional Hospital are AV-recorded are collected and saved for analyzing with consent from all participant.
2. Develop a scoring tool to rate clinical performance in OES. 12 Ekspert Senior Obstetricians from different maternity units in Britain, Norway, Sweden, Denmark and Iceland volunteered to join the Delphi panel and develop a clinical performance tool.
3. Rate clinical performance. Using the developed tool in 2) to rate live teams
4. Rate NTS Recording of teams will be rated by the validated list: Assessment of Obstetric Team Performance with the validated tool from Pamela Morgan: AOTP. Furthermore important observations will be code. Video assessments is planned for 2016-2018
5. Explore the association between clinical performance and NTS in OES. Results from 3) and 4) will be compared.

Discussion:

We expect that this study will add to the knowledge of NTS and the effect on clinical performance in OES.

ELIGIBILITY:
Inclusion Criteria:

Video recordings of emergency situations in simulation aswell live will include management of every day situations as well as rare emergencies, with the inclusion criteria of obstetric teamwork: >2 healthcare personal present and one of them an obstetrician. The five situations in are study are the following:

1. Eclampsia,
2. Post-partum haemorrhage,
3. New -born resuscitation (Apgar ≤ 7/5 min),
4. Shoulder dystocia and
5. Instrumental delivery. The situation can be included if a video recording is capture of the event and all participant in the video have given informed consent.

Exclusion Criteria:

Absent informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the study will include working staff (junior and senior doctors, midwifes and other health personal) in the maternity wards of two hospitals in Central Region Denmark: Horsens Regional Hospital and Aarhus University Hospital, Skejby. Video recording in simulation as well in reality will take place in both hospitals. Approximately 200 different teams each of 3-5 persons will participate in the study. In the live emergency scenarios
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 15. october 2014 - 20. May 2016
  Clinical performance is assessed by video raters, using a checklist TeamOBS-tool

SECONDARY OUTCOMES:
Blood loss | 15. october 2014 - 20. May 2016
  Blood loss measured and verbalized by the emergency team.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, MD.PHD, Study Chair — University of Aarhus; Ole Kierkegaard, MD, Principal Investigator — Horsens Hospital
Locations (2):
- Denmark (2):
  - Aarhus University hospital Skejby, Aarhus, DK
  - Horsens Hospital, Horsens, DK

IPD SHARING:
Plan to Share IPD: Undecided